CLINICAL TRIAL: NCT04402684
Title: Influenza Vaccination in Patients Living With HIV in the Northern Region: An Observational Monocentre Study of Blankets, Modalities, Drivers and Brakes
Brief Title: Influenza Vaccination in Patients Living With HIV in the Northern Region
Acronym: VACCIGRIPPE
Status: Completed | Type: Observational
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH_2020_5
Record Dates: First submitted 2020-04-17; First posted 2020-05-27 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anyone living with the Human Immunodeficiency Virus (HIV) has an indication for annual influenza vaccination. (Vaccination schedule and vaccination recommendations 2019). Influenza is a viral infection that has a significant impact on the health care system. However, vaccination coverage in France is still insufficient with regard to the objectives set at 75% by the WHO and the European Commission. For the 2019-2020 seasonal influenza vaccination campaign, flu vaccination by volunteer pharmacists has become possible throughout the country. Studies that have estimated vaccination coverage among HIV-positive populations are rare and show very low rates.

DETAILED DESCRIPTION:
Cross-sectional study via a self-questionnaire given to all HIV-infected patients coming for a scheduled consultation as part of their HIV follow-up in the spring of 2020. Non-opposition letter given to the patient. Collection of data a posteriori from the medical file recorded in the eNadis patient file.

ELIGIBILITY:
Inclusion Criteria:

* Any adult person living with HIV presenting for a follow-up consultation in the spring of 2020
* People who do not read French may participate if they wish with the help of a medical or paramedical staff member.
* Patient did not object

Exclusion Criteria:

* Minor patients
* Major under guardianship, curatorship, protected person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult person living with HIV presenting for a follow-up consultation in the spring of 2020
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
questionnaire influenza vaccine coverage | through study completion, an average of 1 year
  The objective of this questionnaire is to estimate the influenza vaccine coverage among PVVIH followed at the Tourcoing Hospital Center.

SECONDARY OUTCOMES:
modalities of influenza vaccination | through study completion, an average of 1 year
  To identify the modalities of influenza vaccination when it is carried out
the drivers and disincentives to influenza vaccination | through study completion, an average of 1 year
  Estimate from patient reports the drivers and disincentives to influenza vaccination in a specific risk population.

CONTACTS AND LOCATIONS:
Overall Officials: Macha TETART, MD, Principal Investigator — CH TOURCOING
Locations (1):
- CH Tourcoing, Tourcoing, France

IPD SHARING:
Plan to Share IPD: No